CLINICAL TRIAL: NCT00905437
Title: Randomized Double-Blind, Multi-Center Study Of Efficacy And Tolerability Of Pregabalin Versus Placebo As An Adjunct To Standard Of Care For Perioperative Management Of Patients Undergoing Total Hip Arthroplasty
Brief Title: Study To Investigate The Effectiveness Of Pregabalin For Management Of Patients Undergoing Total Hip Replacement
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Study was terminated on May 24th 2012 due to a slow recruitment rate. The study was not terminated for reasons of safety or efficacy.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: A0081229
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pain, Perioperative
Keywords: perioperative; pregabalin; total hip replacement; post-operative pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo as an adjunct to standard of care
  Interventions: Drug: Placebo
- Pregabalin (Active Comparator): Pregabalin as an adjunct to standard of care
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Placebo — Placebo as an adjunct to standard of care
  Arms: Placebo
Drug: Pregabalin — 75 mg BD for 14 days
  Arms: Pregabalin

SUMMARY:
The purpose of this study is the investigate if pregabalin started a day before surgery and continued for 14 days post-operatively can reduce post-operative pain, relieve pre- and post-operative anxiety and sleep disturbances.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing a routine (i.e., expected to be uncomplicated) total primary or secondary hip replacement surgery performed under a standardized regimen of spinal anesthesia, and is expected to experience moderate to severe post-surgical pain in the absence of post-operative analgesia

Exclusion Criteria:

* The patient is undergoing a revision to a previous hip replacement procedure, hip replacement procedure further to a road traffic accident with multiple injuries, or a procedure expected to last longer than 4 hours
* The patient has a history of uncontrolled chronic disease or a concurrent clinically significant illness or medical condition, which in the Investigator's opinion, would contraindicate study participation or confound interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kanpur, Uttar Pradesh
  - Pfizer Investigational Site, Kolkata, West Bengal
  - Pfizer Investigational Site, New Delhi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081229&StudyName=Study%20To%20Investigate%20The%20Effectiveness%20Of%20Pregabalin%20For%20Management%20Of%20Patients%20Undergoing%20Total%20Hip%20Replacement%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Pregabalin 75 milligram (mg) capsule orally twice daily for 14 days.
- Placebo: Placebo matched to pregabalin 75 mg capsule orally twice daily for 14 days.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 35 | 37
Completed | 27 | 27
Not Completed | 8 | 10
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13.5) | 48.9 (13.3) | 48.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain on Movement Score
Description: Mean pain on movement score was defined as the mean of the pain on movement score over Days 1 to 5 post-surgery. Pain experienced by participant during passive flexion through 90 degree and passive abduction through 30 degree at operated hip joint was evaluated on a scale of 0 to 10 where, 0= no pain and 10= worst possible pain.
Time Frame: Every 12 hours from Day 1 to Day 5 post-surgery
Population: Modified Intent to Treat (MITT) population included all randomized participants who had at least taken pre-surgery study medication and had no surgical complications. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 27 | 30
Units on a scale | 4.0 (0.23) | 3.9 (0.26)

2. Secondary Outcome: Mean Daily Pain Score
Description: Mean daily pain score was defined as the mean of daily pain score over Days 1 to 7 and Days 8 to 14 post-surgery. Daily Pain Rating Scale (DPRS): participant rated 11-point Likert scale ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicates greater level of pain.
Time Frame: Day 1 to Day 7, Day 8 to Day 14 post-surgery
Population: MITT population included all randomized participants who had at least taken pre-surgery study medication and had no surgical complications. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure. 'n' signifies participants who were evaluable for this measure at specified time-point for each arm.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 27 | 30
Units on a scale
  Days 1 to 7 (n=27,30) | 2.6 (0.23) | 2.6 (0.24)
  Days 8 to 14 (n=26,27) | 1.8 (0.25) | 1.4 (0.25)

3. Secondary Outcome: Mean Daily Sleep Interference Score
Description: Mean daily sleep interference score was defined as the mean of daily sleep interference numeric rating scale (NRS) score over Days 1 to 5 post-surgery. Daily Sleep Interference Scale (DSIS): participant rated pain during past 24-hour period on NRS ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep). Higher score indicates a greater level of sleep disturbance. Self-assessment performed daily on awakening prior to taking study medication.
Time Frame: Day 1 to Day 5 post-surgery
Population: MITT population included all randomized participants who had at least taken pre-surgery study medication and had no surgical complications. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 27 | 30
Units on a scale | 2.6 (0.34) | 3.1 (0.29)

4. Secondary Outcome: Mean Anxiety Visual Analogue Scale (A-VAS)
Description: Mean anxiety visual analogue scale (VAS) was defined as the mean of VAS score on the day of surgery and over Days 1 to 5 post-surgery. Participants measured their degree of anxiety over past 24 hours on a VAS of 0 to 100, where 0 = not at all anxious to 100 = extremely anxious.
Time Frame: Day 0 to Day 5 post-surgery
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 36
Units on a scale | 23.3 (3.33) | 24.7 (2.88)

5. Secondary Outcome: Time to Mobilization After Surgery
Description: Participant was encouraged each day (from Day 3) to attempt walking depending upon the degree of pain on standing. The first day on which the participant was able to walk for 5 steps was the day of mobilization. Median time to mobilization (in hours) was calculated till the day of mobilization.
Time Frame: Day 1 to Day 5 post-surgery
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 33 | 35
hours | 72.500 [51.250 to 76.167] | 52.417 [46.750 to 73.250]

6. Secondary Outcome: Number of Participants With Rescue Medication Usage
Description: Rescue medications were used for participants with moderate or severe resting pain. Fentanyl injection (25 microgram [mcg] intravenous bolus to a maximum dose of 3 milliliter/day), paracetamol tablet (15 milligram/kilogram orally to a maximum dose of 45 milligram/kilogram/day) were used as rescue medications.
Time Frame: Day 0 to Day 6 post-surgery
Population: MITT population included all randomized participants who had at least taken pre-surgery study medication and had no surgical complications.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 33 | 36
participants | 17 | 25

7. Secondary Outcome: Number of Participants With Neuropathic Pain
Description: ID Pain questionnaire was used to assess neuropathic pain. 6 items questionnaire, did pain feel like: (1)pins and needles (2)hot/burning (3)numb (4)electrical shocks (5)is pain made worse with touch of clothing or bed sheets (6)is pain limited to your joints. "Yes" response to questions 1-5 were scored as 1, while a "yes" response to question 6 was scored as -1. "No" response were scored as 0. Overall score range -1 to 5.Higher score more indicative of pain with a neuropathic component. Number of participants with score 2 or more (which indicated nerve pain) were reported.
Time Frame: Day 90, Day 180 post-surgery
Population: Data was not analyzed as the intended sample size was not met, and the reported numbers from the final set were not sufficient for a meaningful analysis.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/35 | 0/37
Other Adverse Events (participants affected / at risk) | 23/35 | 22/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=35) | Placebo (N=37)
Oxygen saturation decreased (Investigations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=35) | Placebo (N=37)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 16 | 10
Drug hypersensitivity (Immune system disorders) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Urinary retention postoperative (Infections and infestations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
As the enrollment rate was very low, the study was prematurely terminated. The number of enrolled participants was too low for meaningful formal statistical conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.